CLINICAL TRIAL: NCT01804959
Title: A Proof-of-concept Double-blind Randomized Placebo-controlled Trial of Probiotics in Systemic Sclerosis Associated Gastrointestinal Disease
Brief Title: Clinical Trial of Probiotics in Systemic Sclerosis Associated Gastrointestinal Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AL-SScGI
Record Dates: First submitted 2013-03-03; First posted 2013-03-05 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active vs Placebo (Placebo Comparator): In phase I, subjects will be randomized into either the Vivomixx probiotics or placebo arm of the study at a 1:1 ratio. All randomized subjects will receive probiotics (4 sachets/ day or 1800 billion bacteria/day) or placebo (4 placebo sachets/day) for the first 60 days.
  Interventions: Dietary Supplement: Vivomixx probiotics
- 60 days of Active vs 120 days of Active (Active Comparator): In phase II, subjects from both arms in phase I will receive Vivomixx probiotics 4 sachets/ day for another 60 days. Comparison will be made between the arm receiving 60 days of Vivomixx probiotics vs 120 days of Vivomixx probiotics
  Interventions: Dietary Supplement: Vivomixx probiotics

INTERVENTIONS:
Dietary Supplement: Vivomixx probiotics

SUMMARY:
SSc-associated gastrointestinal (GI) involvement is common, with no effective treatment. Probiotics may have beneficial effects on symptoms as supported by one small open-label study (n=10) that demonstrated decreased bloating symptoms in SSc patients after 2 months of probiotics. This study aims to determine (i) whether 60 days of Vivomixx probiotics result in greater GI symptom improvement than placebo in SSc outpatients, assessed using an interview-administered 34-item Gastrointestinal Tract (GIT) questionnaire and (ii) whether 60 days versus 120 days of probiotics result in greater GI symptom improvement in SSc outpatients, assessed using the GIT questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* SSc that fulfills the American College of Rheumatology (ACR, 1990) classification criteria or the proposed European League Against Rheumatism (EULAR) criteria for very early diagnosis of systemic sclerosis.
* SSc overlap syndromes (ie SSc occurring in overlap with other connective tissue diseases)
* SSc-associated GI symptoms (heartburn, dysphagia, vomiting, bloating/distension, faecal soilage, diarrhoea, constipation) not due to other causes as determined by clinical evaluation, with a total GIT score of at least 0.10
* Stable doses of immunosuppressive treatment, corticosteroids, and GI medications for 30 days.

Exclusion Criteria:

* On anti-biotics or probiotics within the last 30 days
* Current serious infections requiring hospitalization
* Long-term indwelling catheter, including patients on total parenteral nutrition
* Females who are lactating or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2017-11 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
mean difference between probiotics group versus placebo group in gastrointestinal change score from baseline to day 60 of treatment. | After 60 days of either placebo treatment or active drug treatment

SECONDARY OUTCOMES:
mean difference between 60 days of probiotics versus 120 days of probiotics in gastrointestinal change score from baseline to day 120 of treatment. | After 120 days of placebo treatment or active drug treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Low AHL, Teng GG, Pettersson S, de Sessions PF, Ho EXP, Fan Q, Chu CW, Law AHN, Santosa A, Lim AYN, Wang YT, Haaland B, Thumboo J. A double-blind randomized placebo-controlled trial of probiotics in systemic sclerosis associated gastrointestinal disease. Semin Arthritis Rheum. 2019 Dec;49(3):411-419. doi: 10.1016/j.semarthrit.2019.05.006. Epub 2019 May 23. PMID 31208714